CLINICAL TRIAL: NCT01414699
Title: The Influence of Dietary Variety and Course Sequence on Fruit Intake in Preschool-Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 8585B
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Caloric Intake
Keywords: dietary variety; course sequence; preschool; child feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- One-Course, Variety (Active Comparator): Participants will receive a snack in one course with a variety of fruit.
  Interventions: Behavioral: Variety
- Two-Course, Variety (Active Comparator): Participants will receive a snack in two courses with a variety of fruit.
  Interventions: Behavioral: Variety
- One-course, Non-Variety (Active Comparator): Participants will receive a snack in one course with no variety of fruit.
  Interventions: Behavioral: Non-Variety
- Two-Course, Non-Variety (Active Comparator): Participants will receive a snack in two courses with no variety of fruit.
  Interventions: Behavioral: Non-Variety

INTERVENTIONS:
Behavioral: Variety — These conditions will have snack served with an increase of fruit variety.
  Arms: One-Course, Variety; Two-Course, Variety
Behavioral: Non-Variety — These conditions will receive a snack without a variety of fruit.
  Arms: One-course, Non-Variety; Two-Course, Non-Variety

SUMMARY:
The purpose of this study is to determine the extent to which manipulation of dietary variety and course sequence affects fruit intake and overall energy intake in preschool-aged children.

DETAILED DESCRIPTION:
In the past two decades overweight and obesity rates in children (ages 2-19) have risen from 5% to 17%, with toddlers (ages 2-5) at 10%. Among children and adolescents the consumption of low-energy-dense foods, such as fruit and vegetables (F&Vs), remain below current recommendations. Therefore, strategies to increase low-energy-dense F&V intake and decrease high-energy-dense food intake aimed at young children are essential. Antecedents, or cues, can trigger eating. Therefore, manipulating food presentation can be utilized to produce certain behaviors. Dietary variety and course sequence are two examples of this relationship. It has been well established that high dietary variety leads to greater consumption patterns compared to low DV diets in adults. High DV has only been tested with problematic foods, and not with the goal of increasing F&V intake. Additionally, serving a first course meal can act as a preload to decrease intake of the second course entrée. Dietary variety and course sequence manipulations have been experimentally tested with caloric intake goals but never with the goal of increasing F&V intake. Therefore, the purpose of this study is to determine the extent to which manipulation of dietary variety and course sequence affects fruit intake and overall energy intake in preschool-aged children.

ELIGIBILITY:
Inclusion Criteria:

* All children that are ≥3 years of age enrolled in the ELC preschool with parental consent can participate.
* Eligible children must also like applesauce, peaches and cheese cubes, and be able to consume foods with a spoon.

Exclusion Criteria:

* Children allergic to applesauce, peaches, or chocolate pudding or who are lactose-intolerant will not be included in the study.
* Did not attend all feeding sessions.
* Did not consume more than 5 grams from any of the foods on an occasion.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total grams of snack consumed. | 4 weeks
  Total grams of snack consumed by participants over the 4-week study (with 1 snack per week) period will be determined by subtracting pre- and post-consumption weight of the snack provided.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — University of Tennessee, Knoxville; Chelsi C Cardoso, BS, Principal Investigator — University of Tennessee, Knoxville
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this study is being conducted. — http://heal.utk.edu